CLINICAL TRIAL: NCT00587093
Title: Multicenter Trial on Utility and Impact of Computed Tomography and Serum CA-125 in Management of Newly Diagnosed Ovarian Cancer
Brief Title: A Multicenter Trial On The Utility and Impact Of Computed Tomography and Serum CA-125 In the Management of Newly Diagnosed Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Johns Hopkins University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-048; NCT00502151 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Cancer
Keywords: Newly diagnosed; CA 125; CT scan; 01-048
MeSH Terms: conditions — Ovarian Neoplasms | interventions — CA-125 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): CT scan and CA-125
  Interventions: Other: CA 125 and CT scan

INTERVENTIONS:
Other: CA 125 and CT scan — Within 14 days prior to surgery serum for CA125 will be obtained. The patient will also undergo a CT scan of the abdomen and pelvis with oral and intravenous contrast within 35 days prior to the procedure.

SUMMARY:
The purpose of the research is to determine if blood tests and a CT scan done before surgery can predict how successful the surgery will be. In patients who have cancer of the ovary that has spread, it is hoped that the CT scan will be able to identify the various places where the cancer has spread so that additional surgeons can be available to help with the surgical procedure.

If you have confirmed stage 3 or 4 ovarian, fallopian tube, or primary peritoneal cancer, you may undergo a CT scan of the abdomen and pelvis after the surgery to compare how much cancer the surgeon thought was left after surgery to what is seen on CT scan. A CT scan of the chest will be done if your physician thinks it is necessary.

DETAILED DESCRIPTION:
This study is designed to assess the utility and impact of computed tomography (CT)scanning of the abdomen and pelvis and preoperative serum CA-125 levels in the management of patients undergoing surgery for presumed ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 years of age undergoing surgery for presumed ovarian, fallopian tube, or primary peritoneal cancer.
* Patients must be medically and physically able to undergo general anesthesia and possible tumor debulking.
* Patients must read and sign informed consent form after the nature of the study has been fully explained.

Exclusion Criteria:

* Presence of clinically significant disease, allergy, or other disorder precluding the ability to safely perform CT scan of the abdomen and pelvis with oral and intravenous contrast.
* Vulnerable patients (minors, mentally retarded patients, prisoners, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2001-07 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of preoperative CT scan of the abdomen and pelvis in predicting optimal primary cytoreduction in advanced ovarian cancer. | 7 - 35 days postop stage 3 or 4 disease CTscan have

SECONDARY OUTCOMES:
To evaluate the ability of preoperative serum CA-125 to predict optimal primary cytoreduction of advanced ovarian cancer. | Within 14 days prior to surgery
To develop preoperative CT scan of the abdomen and pelvis and/or tumor marker criteria for ovarian cancer non-resectability (sub-optimal tumor cytoreduction). | 3 years
To determine the ability of preoperative CT scan of the abdomen and pelvis to provide useful information that will impact on surgical planning. | 3 years
To compare the intraoperative assessment of residual disease to that found on postoperative CT scan of the abdomen and pelvis, if scans are available for review. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org